CLINICAL TRIAL: NCT04561947
Title: Clinical Evaluation of the Treatment of Multiple Gingival Recessions with Connective Tissue Graft or Concentrated Growth Factor Membrane Using Tunnel Technique: a Randomized Controlled Clinical Trial
Brief Title: Treatment of Gingival Recessions with Connective Tissue or Concentrated Growth Factor Membrane Using Tunnel Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Umut BALLI, Associate professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-82-09/08
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2020-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TT+CTG (Active Comparator): The combined connective tissue graft (CTG) with tunnel technique (TT)
  Interventions: Procedure: Tunnel technique; Procedure: Connective tissue graft
- TT+CGF (Experimental): The combined concentrated growth factor (CGF) membrane with tunnel technique (TT)
  Interventions: Procedure: Tunnel technique; Other: Concentrated growth factor membrane

INTERVENTIONS:
Procedure: Tunnel technique — After local anesthesia, the exposed root surfaces were mechanically treated with curettes. A tunnelling knives were used to prepare a split-thickness flap and create a continuous tunnel in the buccal soft tissues, following the intrasulcular incision with a #69 microblade. Split-thickness flap preparation was performed to beyond the mucogingival junction with supraperiosteal dissection by placing the tunneling knives to the soft tissue. This process was repeated by entering through the sulcus of each tooth. After the elevation of the flap, a papilla elevator placed under the flap was entered through the sulcus to mobilize the papilla, the periosteum at the base of the papilla was cut, and the full-thickness flap was elevated.
Procedure: Connective tissue graft — CTG was harvested using the de-epithelialized connective tissue graft technique. The epithelial tissue on the outer surface of the graft was removed with a 15 blade and a 1-mm-thick graft was obtained.
  Arms: TT+CTG
Other: Concentrated growth factor membrane — Intravenous blood samples were collected in without anticoagulant 10-mL tubes and immediately centrifuged in a CGF centrifuge machine using a program with the following features: 30 ̋ acceleration, 2 min at 2700 rpm, 4 min at 2400 rpm, 4 min at 2700 rpm, 3 min at 3000 rpm, and 36 ̋ deceleration and stop. After centrifugation, four layers were formed in the tube: the serum layer at the top, the second buffy coat layer, the third CGF layer containing GF and unipotent stem cells, and the red blood cell layer at the bottom. The resulting CGF was removed from the tube and separated from the red blood cell layer using microsurgical scissors.
  Arms: TT+CGF

SUMMARY:
This randomized controlled clinical study aimed to evaluate the success of the combination of tunnel technique and concentrated growth factor membrane for root coverage in treating multiple gingival recessions and compare with the gold standard connective tissue graft.

DETAILED DESCRIPTION:
The study included 108 defects in 40 patients with Miller Class I and II gingival recession. Gingival recession defects were randomly divided into two groups. Tunnel technique + connective tissue graft was applied to 20 patients in the control group (51 defects) and tunnel technique + concentrated growth factor membrane was applied to 20 patients in the test group (57 defects). The results at baseline and 6 months were evaluated for the following clinical parameters: Mean root coverage, complete root coverage, probing depth, clinical attachment level, gingival recession depth, gingival recession width, keratinized tissue width and gingival thickness.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* periodontally and systemically healthy
* presence of Miller I or II class gingival recession defect in at least two teeth on the buccal aspect of incisors, canine and premolar teeth (≥ 2 mm in depth)
* gingival thickness ≥ 0.8 mm 2 mm apical to the gingival margin
* presence of identifiable cementoenamel junction (CEJ) (step ≤1 mm at the CEJ level and/or presence of a root irregularity/abrasion with identifiable CEJ was accepted
* full-mouth plaque score (FMPS) ≤20%.

Exclusion Criteria:

* smoking
* contraindications for surgical periodontal treatment
* presence of recession defects associated caries, restoration and furcation problems
* use of systemic antibiotics for any reason in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | Six months
  Change from baseline in percentage of complete root coverage at 6th months.

SECONDARY OUTCOMES:
Mean root coverage | Six months
  Change from baseline in percentage of root coverage at 6th months.
Probing depth | Six months
  Change from baseline in probing depth at 6th months. The distance between the sulcus base and the gingival margin the midbuccal aspect of the teeth
Clinical attachment level | Six months
  The changes in clinical attachment level after 6th months. Distance between the sulcus base and the CEJ in the midbuccal aspect of the teeth
Gingival recession depth | Six months
  The changes in gingival recession depth after 6th months. Distance between the gingival margin at the deepest point of recession
Gingival recession width | Six months
  The changes in gingival recession width after 6th months. Horizontal distance between the mesial and distal margin of the recession defect at the CEJ
Keratinized tissue width | Six months
  The changes in keratinized tissue width after 6th months. Distance between the gingival margin and the mucogingival junction
Gingival thickness | Six months
  The changes in gingival thickness after 6th months. Measured midbuccally from 2 mm apical to the gingival margin with a No: 20 endodontic spreader

CONTACTS AND LOCATIONS:
Overall Officials: Birsen KORKMAZ, assis. Prof., Principal Investigator — birsenkorkmaz91@gmail.com; Umut BALLI, Assoc. Prof., Study Director — ZBEU.
Locations (1):
- Bulent Ecevit U., Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Korkmaz B, Balli U. Clinical evaluation of the treatment of multiple gingival recessions with connective tissue graft or concentrated growth factor using tunnel technique: a randomized controlled clinical trial. Clin Oral Investig. 2021 Nov;25(11):6347-6356. doi: 10.1007/s00784-021-03935-3. Epub 2021 Apr 8. PMID 33830339